CLINICAL TRIAL: NCT06118021
Title: A Randomized, Double-blind, Placebo-controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of HS-20094 in Overweight and Obese Subjects
Brief Title: A Study of HS-20094 Evaluating Weight Loss in Obese and Overweight Chinese Subjects
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-20094-202
Record Dates: First submitted 2023-10-17; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HS-20094 5mg (Experimental): Drug: HS-20094 administered subcutaneously (SC) once a week. Drug: Placebo administered subcutaneously (SC) once a week.
  Interventions: Drug: HS-20094; Drug: Placebo
- HS-20094 10mg (Experimental): Drug: HS-20094 administered subcutaneously (SC) once a week. Drug: Placebo administered subcutaneously (SC) once a week.
  Interventions: Drug: HS-20094; Drug: Placebo
- HS-20094 15mg (Experimental): Drug: HS-20094 administered subcutaneously (SC) once a week. Drug: Placebo administered subcutaneously (SC) once a week.
  Interventions: Drug: HS-20094; Drug: Placebo
- HS-20094 20mg (Experimental): Drug: HS-20094 administered subcutaneously (SC) once a week. Drug: Placebo administered subcutaneously (SC) once a week.
  Interventions: Drug: HS-20094; Drug: Placebo

INTERVENTIONS:
Drug: HS-20094 — Administered SC
  Other Names: HS-20094 injection
Drug: Placebo — Administered SC
  Other Names: Placebo injection

SUMMARY:
This is a study of HS-20094 in participants with overweight and obesity. The main purpose is to learn more about how HS-20094 affects body weight. The study period including 4-12 weeks dose titration and 12-20 weeks maintain treatment and 6 weeks follow up.

DETAILED DESCRIPTION:
This is a phase 2, double-blind, randomised, placebo-controlled trial to assess the efficacy of HS-20094 in Chinese subjects with overweight or obesity. We enrolled adults (aged 18-65 years, both inclusive) with overweight (body-mass index [BMI] ≥24 kg/m2) accompanied by at least one obesity-related comorbidity or obesity (BMI ≥28 kg/m2) from over 10 hospitals in China. Eligible participants were randomly assigned (4:1) within each cohort by using an interactive web-response system to receive once-weekly subcutaneous HS-20094 or placebo for 24 weeks in one of the 4 cohorts below：the 5 mg cohort (5 mg weeks 1-24) ，the 10 mg cohort（5 mg weeks 1-4，10 mg weeks 5-24），the 15 mg cohort（5 mg weeks 1-4，10 mg weeks 5-8,15 mg weeks 9-24），the 20 mg cohort（5 mg weeks 1-4，10 mg weeks 5-8，15 mg weeks 9-12，20 mg weeks 13-24）. The participants, investigators, study site personnel involved in treating and assessing participants in each cohort and sponsor personnel were masked to treatment allocation. The primary endpoints were the percent change in bodyweight from baseline and bodyweight reduction of 5% or higher. The secondary outcomes included the change from baseline to week 24 in waist circumference and BMI.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects,18-65 years of age at the time of signing informed consent.
2. BMI≥28.0kg/m2 or 24≤BMI<28.0 kg/ m2 with at least 1 weight-related comorbidity at screening visit.
3. Diet and exercise control for at least 3 months before screening visit,and less than 5 kg self-reported change within the last 3 months.

Exclusion Criteria:

* 1. Presence of-clinically significant lab or ECG results that may affect the evaluation of the efficacy or safety of the study drug at screening visit.

  2. poor-controlled hypertension. 3. PHQ-9 score≥15. 4. Medical history or illness that affects your weight. 5. Use of any medication or treatment that may have caused significant weight change within 3 months.

  6. History of bariatric surgery. 7. History of diabetes. 8. Acute infection, acute trauma, or medium to large surgery within 1 month prior to screening.

  9. History of acute cardiovascular and cerebrovascular diseases within 6 months prior to screening.

  10. Any organ-system malignancies developed within 5 years except for cured local basal cell cancer of the skin and in-situ cancer of the cervix.

  11. Confirmed or suspected depression, bipolar disorder, suicidal tendencies, schizophrenia, or other serious mental illness.

  12. History of alcohol and/or substance abuse or drug abuse within 1 year prior to screening.

  13. Participation in other clinical trials for any weight-loss indication within 3 months prior to screening, or participation in other clinical trials for any drug or medical device within 1 month prior to screening.

  14. Known or suspected hypersensitivity to trial product(s)or related products. 15. Female who is pregnant,breast-feeding or intends to become pregnant or is of childbearing potential and not using an adequate contraceptive method.

  16. Researchers and relevant staff of the research Centre or other people directly involved in the implementation of the programme,and their immediate family members.

  17. In the judgment of the investigator,there are circumstances that affect the safety of the subject or any other interference with the evaluation of the test results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-10-16 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Weight | From Week 0 to Week 24
  Percent Change from Baseline in Body Weight

SECONDARY OUTCOMES:
Number of AEs During the Trial | From Week 0 to Week 24
  Safety
Change from Baseline in Patient Health Questionnaire-9 (PHQ-9) | From Week 0 to Week 24
Change from Baseline in Columbia Suicide Severity Rating scale ( C-SSRS) | From Week 0 to Week 24
12-lead electrocardiogram (ECG) parameters: PR, R-R, QRS and QTcF (average) | From Week 0 to Week 24
Change from baseline in waist circumference after 24 weeks of treatment | From Week 0 to Week 24
Change from baseline in BMI after 24 weeks of treatment | From Week 0 to Week 24
Change from baseline in blood pressure after 24 weeks of treatment | From Week 0 to Week 24
Change from baseline in total cholesterol after 24 weeks of treatment | From Week 0 to Week 24
Change from baseline in fasting plasma glucose(FPG)after 24 weeks of treatment | From Week 0 to Week 24

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - the Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang